CLINICAL TRIAL: NCT06698250
Title: Phase II Trial of Zanzalintinib (XL-092) in Combination With Durvalumab Plus Tremelimumab in Unresectable Hepatocellular Carcinoma (ZENOBIA)
Brief Title: Zanzalintinib (XL-092) Plus Durvalumab and Tremelimumab in Unresectable Hepatocellular Carcinoma (ZENOBIA)
Acronym: ZENOBIA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anwaar Saeed (Other)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor-Investigator, Anwaar Saeed, Associate Professor & Chief of GI Medical Oncology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC 23-116; XL092- IST207 (Other: Exelixis Protocol Number)
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: tyrosine kinase inhibitor (TKI); vascular endothelial growth factor (VEGF); AXL receptor tyrosine kinase (AXL); Programmed death-1/programmed death ligand-1 (PD-1/PD-L1)
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Safety Lead-in - Zanzalintinib (XL-092) + Tremelimumab (IV) + Durvalumab (IV) (Experimental): Safety Lead-in: XL-092: The first dose level (dose level 0) will follow the rolling 6 design*. The participants enrolled in this study part will receive one cycle of XL-092 60 mg orally (PO) daily plus durvalumab 1500 mg intravenously (IV) every 28 days + tremelimumab 300 mg IV once. In cycle 2 and subsequent cycles, participants will receive XL-092 60 mg orally (PO) daily and durvalumab 1500mg IV every 28-day cycles. DLT period will be 28 days.
  One level dose reduction will be pursued based DLT read of the dose level 0 participants.
  For dose level -1, XL-092 will be used at 40mg daily dosing, in combo with the same flat dosings for Durvalumab and Tremelimumab. Safety lead in will be 6-12 patients.
  Interventions: Drug: Zanzalintinib; Drug: Durvalumab; Drug: Tremelimumab
- Zanzalintinib (XL-092) + Tremelimumab (IV) + Durvalumab (IV) (Begin First Cyle Zanzalintinib) (Active Comparator): Phase 2: One cycle of XL-092 RP2D PO daily + durvalumab 1500 mg intravenously (IV) every 28 days + tremelimumab 300 mg IV once. XL- 092 RP2D daily and durvalumab will then be continued every 28 days cycles until discontinuation due to disease progression, intolerability, or withdrawal of consent.
  Interventions: Drug: Zanzalintinib; Drug: Durvalumab; Drug: Tremelimumab
- Zanzalintinib (XL-092) + Durvalumab (IV) + Tremelimumab (IV) (Begin Second Cyle Zanzalintinib) (Active Comparator): Phase 2: One cycle of durvalumab 1500 mg IV + tremelimumab 300 mg IV once followed by XL-092 RP2D mg PO Daily + durvalumab 1500 mg IV every 28 days until discontinuation due to disease progression, intolerability, or withdrawal of consent.
  Interventions: Drug: Zanzalintinib; Drug: Durvalumab; Drug: Tremelimumab

INTERVENTIONS:
Drug: Zanzalintinib — Next generation tyrosine kinase inhibitor (TKI) with the target inhibition proﬁle identical to cabozantinib but with a superior pharmacokinetic proﬁle.
  Other Names: XL-092
Drug: Durvalumab — Durvalumab is a human immunoglobulin G1 kappa (IgG1κ) monoclonal antibody that blocks the interaction of programmed cell death ligand 1 (PD-L1) with the PD-1 (CD279)
  Other Names: Imfinzi
Drug: Tremelimumab — Tremelimumab is a fully human monoclonal antibody used for the treatment of hepatocellular carcinoma designed to attach to and block CTLA-4, a protein that controls the activity of T cells
  Other Names: Imjudo

SUMMARY:
This study will investigate if modulating the tumor microenvironment with biologic agents like XL-092 will have synergistic eﬀect when combined with checkpoint based immunotherapeutic treatment of patients with hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
Zanzalintinib (XL-092) is a next generation tyrosine kinase inhibitor (TKI) with the target inhibition proﬁle identical to cabozantinib but with a superior pharmacokinetic proﬁle. As cabozantinib targets multiple tyrosine kinases, including vascular endothelial growth factor receptor (VEGFR), MET proto-oncogene, receptor tyrosine kinase (MET), and AXL receptor tyrosine kinase (AXL), and has been reported to show immunomodulatory properties that may counteract tumor-induced immunosuppression, XL-092 is expected to have similar immune modulatory activity, providing a rationale for combining it with PD-1 or PD-L1 inhibitors. This study asserts the belief that modulating the tumor microenvironment with biologic agents like XL-092 will have synergistic eﬀect when combined with checkpoint based immunotherapeutics like durvalumab and tremelimumab in patients with hepatocellular carcinoma (HCC). There will be a Safety lead-in to deﬁne the Recommended Phase 2 Dose (RP2D) that will enroll 6-12 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have unresectable hepatocellular carcinoma.
2. Patients must be treatment naïve for systemic therapy in the unresectable setting.
3. ≥ 18 years and ECOG performance status 0-1
4. Recovery to baseline or ≤ Grade 1 severity (CTCAE v5) from adverse events (AEs), unless AE(s) are clinically nonsigniﬁcant and/or stable on supportive therapy (e.g., physiological replacement of mineralocorticosteroid).
5. Adequate organ and marrow function, based upon meeting all of the following laboratory criteria within 14 days before ﬁrst dose of study treatment.
6. Urine protein-to-creatinine ratio (UPCR) ≤ 1 mg/mg (≤ 113.2 mg/mmol) creatinine. Tumor tissue fresh biopsies are REQUIRED for ALL study participants at screening/baseline unless an archival tumor tissue block is available and fulﬁlls the criteria

   • Note that PI approval can be obtained if institution is unable to release blocks.
7. Capable of understanding and complying with the protocol requirements and must have signed the informed consent document.
8. Sexually active fertile subjects and their partners must agree to use highly eﬀective method of contraception prior to study entry, during the course of the study, and for the following durations after the last dose of treatment (whichever is later). An additional contraceptive method, such as a barrier method (e.g., condom), is required. In addition, men must agree not to donate sperm and women must agree not to donate eggs (ova, oocyte) for the purpose of reproduction during these same periods.
9. Female subjects of childbearing potential must not be pregnant at screening. Female subjects are considered to be of childbearing potential unless permanent sterilization or documented postmenopausal status criteria are met.

Exclusion Criteria:

1. Prior treatment with XL092, or PD-1/PD-L1 or CTLA-4 inhibitors.
2. Receipt of any type of small molecule kinase inhibitor such as cabozantinib or other MET or Dual MET/HGF monoclonal antibodies or MET/HGF tyrosine kinase inhibitors (TKIs), or any other VEGFR TKIs (including investigational kinase inhibitor) within 2 weeks before ﬁrst dose of study treatment.
3. Receipt of any type of cytotoxic, biologic or other systemic anticancer therapy (including investigational) within 4 weeks before ﬁrst dose of study treatment.
4. Radiation therapy for bone metastasis within 2 weeks, any other radiation therapy within 4 weeks before ﬁrst dose of study treatment. Systemic treatment with radionuclides within 6 weeks before ﬁrst dose of study treatment. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible.
5. Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks before ﬁrst dose of study treatment.

   Note: Subjects with an incidental ﬁnding of an isolated brain lesion < 1 cm in diameter may be eligible after Principal Investigator approval if the lesion is radiographically stable for 4 weeks before ﬁrst dose and does not require treatment per Investigator judgement.

   Note: Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of ﬁrst dose of study treatment.
6. Concomitant anticoagulation with oral anticoagulants (e.g., warfarin and direct thrombin inhibitors) and platelet inhibitors (e.g., clopidogrel).

   Note: Allowed anticoagulants are low-dose aspirin for cardioprotection (per local applicable guidelines) and low molecular weight heparins (LMWH). Therapeutic doses of LMWH are not permitted in subjects with known brain metastases. Subjects treated with therapeutic LMWH must have a screening platelet count > 100,000/μL. Note: Subjects must have discontinued oral anticoagulants within 3 days or 5 half-lives prior to ﬁrst dose of study treatment, whichever is longer.
7. Any complementary medications (e.g., herbal supplements or traditional Chinese medicines) to treat the disease under study within 2 weeks before ﬁrst dose of study treatment.
8. The subject has uncontrolled, signiﬁcant intercurrent or recent illness including, but not limited to, the following conditions:

   a. Cardiovascular disorders: i. Congestive heart failure New York Heart Association Class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias (e.g., ventricular ﬂutter, ventricular ﬁbrillation, Torsades de pointes). ii. Uncontrolled hypertension deﬁned as sustained blood pressure (BP) > 140 mm Hg systolic or > 90 mm Hg diastolic despite optimal antihypertensive treatment. iii. Stroke (including transient ischemic attack [TIA]), myocardial infarction, or other clinically signiﬁcant ischemic event within 12 months before ﬁrst dose of study treatment. iv. Pulmonary embolism (PE) or deep vein thrombosis (DVT) or prior clinically signiﬁcant venous or non-CVA/TIA arterial thromboembolic events within 6 months before to ﬁrst dose of study treatment. Note: Subjects with a diagnosis of DVT within 6 months are allowed if asymptomatic and stable at screening and treated with anticoagulation per standard of care before ﬁrst dose of study treatment. Note: Subjects who don't require prior anticoagulation therapy may be eligible but must be discussed and approved by the Principal Investigator. v. Prior history of myocarditis. b. Gastrointestinal (GI) disorders including those associated with a high risk of perforation or ﬁstula formation: i. Tumors invading the GI-tract from external viscera

   ii. Active peptic ulcer disease, inﬂammatory bowel disease, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, or acute pancreatitis iii. Acute obstruction of the bowel, gastric outlet, or pancreatic or biliary duct within 6 months unless cause of obstruction is deﬁnitively managed and subject is asymptomatic iv. Abdominal ﬁstula, gastrointestinal perforation, bowel obstruction, or intra- abdominal abscess within 6 months before ﬁrst dose. Note: Complete healing of an intra-abdominal abscess must be conﬁrmed before ﬁrst dose of study treatment. v. Known gastric or esophageal varices
9. Clinically signiﬁcant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of signiﬁcant bleeding (e.g., pulmonary hemorrhage) within 12 weeks before ﬁrst dose of study treatment.
10. Cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation.
11. Lesions invading major blood vessel including, but not limited to, inferior vena cava, pulmonary artery, or aorta. Subjects with lesions invading the hepatic portal vasculature are eligible. Note: Subjects with intravascular tumor extension (e.g., tumor thrombus in renal vein or inferior V.

    cava) may be eligible following Principal Investigator approval.
12. Other clinically signiﬁcant disorders that would preclude safe study participation.

    1. Active infection requiring systemic treatment. Note: Prophylactic antibiotic treatment is allowed.
    2. Known infection with acute or chronic hepatitis B or C, known human immunodeﬁciency virus (HIV) or acquired immunodeﬁciency syndrome (AIDS)-related illness.
    3. Known positive test for or suspected infection with SARS-CoV-2 within one month before enrollment. Note: demonstration that the subject has fully recovered from the infection is required to be eligible for enrollment
    4. Serious non-healing wound/ulcer/bone fracture. Note: non-healing wounds or ulcers are permitted if due to tumor-associated skin lesions.
    5. Malabsorption syndrome.
    6. Pharmacologically uncompensated, symptomatic hypothyroidism.
    7. Moderate to severe hepatic impairment (Child-Pugh B or C).
    8. Requirement for hemodialysis or peritoneal dialysis.
    9. History of solid organ or allogeneic stem cell transplant.
13. Major surgery within 8 weeks prior to ﬁrst dose of study treatment. Prior laparoscopic nephrectomy within 4 weeks prior to ﬁrst dose of study treatment. Minor surgery within 10 days before the ﬁrst dose of study treatment. Complete wound healing from major or minor surgery must have occurred at least prior to ﬁrst dose of study treatment.

    Note: Fresh tumor biopsies should be performed at least 7 days before the ﬁrst dose of study treatment. Subjects with clinically relevant ongoing complications from prior surgical procedures, including biopsies, are not eligible.
14. Corrected QT interval calculated by the Fridericia formula (QTcF) > 450 ms for males or > 470 for females within 14 days per electrocardiogram (ECG) before ﬁrst dose of study treatment.

    Note: Triplicate ECG evaluations will be performed and the average of these 3 consecutive results for QTcF will be used to determine eligibility.
15. History of psychiatric illness likely to interfere with ability to comply with protocol requirements or give informed consent.
16. Pregnant or lactating females.
17. Inability to swallow tablets.
18. Previously identiﬁed allergy or hypersensitivity to components of the study treatment formulations.
19. Any other active malignancy or diagnosis of another malignancy within 2 years before ﬁrst dose of study treatment, except for superﬁcial skin cancers, or localized, low grade tumors deemed cured and not treated with systemic therapy. Incidentally diagnosed prostate cancer is allowed if assessed as stage ≤ T2N0M0 and Gleason score ≤ 6.
20. Other conditions, which in the opinion of the Investigator, would compromise the safety of the patient or the patient's ability to complete the study.
21. Any active, known or suspected autoimmune disease requiring long term treatment with immunosuppressive medications. Note: Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
22. Known positive test for tuberculosis infection if supported by clinical or radiographic evidence of disease.
23. History of idiopathic pulmonary ﬁbrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computerized tomography (CT) scan. History of radiation pneumonitis in the radiation ﬁeld (ﬁbrosis) is permitted.
24. Free thyroxine (FT4) outside the laboratory normal reference range. Asymptomatic subjects with FT4 abnormalities can be eligible after Principal Investigator approval.
25. Diagnosis of immunodeﬁciency or is receiving systemic steroid therapy (> 10 mg daily prednisone equivalent) or any other form of immunosuppressive therapy within 2 weeks prior to ﬁrst dose of study treatment. Inhaled, intranasal, intraarticular, and topical corticosteroids and mineralocorticoids are allowed. Note: Adrenal replacement steroid doses > 10 mg daily prednisone equivalent are permitted in the absence of active autoimmune disease. Transient short-term use of higher doses of systemic corticosteroids for allergic conditions (e.g., contrast allergy) is also allowed.
26. Administration of a live, attenuated vaccine within 30 days before ﬁrst dose of study treatment.
27. Documented hepatic encephalopathy (HE) within 6 months before ﬁrst dose of study treatment.
28. Clinically meaningful ascites (i.e., ascites requiring paracentesis or escalation in diuretics) within 6 months before ﬁrst dose of study treatment.
29. Subjects who have received any local anticancer therapy including surgery, regional ablative therapies including thermal ablation, radiofrequency ablation (RFA), Microwave Ablation (MWA) transarterial chemoembolization (TACE), or transarterial radioembolization (TARE) within 28 days prior to ﬁrst dose of study treatment.
30. Child Pugh score > 7.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Recommended phase 2 dose (RP2D) of XL-092 with Durvalumab plus Tremelimumab | Up to 12 months
  Recommended phase 2 dose (RP2D) of XL-092 with Durvalumab plus Tremelimumab will be determined per a Dose Limiting Toxicity period of 28 days during the Safety Lead-in period using CTCAE v5.0 criteria.
Objective Response Rate (ORR) (im RECIST) | Up to 24 months
  Proportion of patients with Complete Response (CR) or Partial Response (PR), per immune modiﬁed RECIST v1.1. Per imRECIST: CR: -100% Change in Sum of Diameters from Baseline (non-target lesion). PR: ≤ -30% change in sum of diameters from baseline.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 24 months
  Proportion of patients with Complete Response (CR) or Partial Response (PR), per RECIST v1.1. CR: Disappearance of all target lesions. Any pathological lymph nodes (target or non-target) with reduction in short axis to <10 mm. PR: ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Rate of Disease Conversion | Up to 12 months
  Proportion of patients able to undergo liver resection or transplantation after completion of treatment.
Disease Control Rate (DCR) | Up to 24 months
  Proportion of patients with Complete Response (CR), Partial Response (PR) or Stable Disease (SD), per immune modiﬁed RECIST v1.1. Per imRECIST: CR: -100% Change in Sum of Diameters from Baseline (non-target lesion). PR: ≤ -30% change in sum of diameters from baseline. SD: >-30% to < +20% change in sum of diameters from baseline.
Progression-free Survival (PFS) | Up to 40 months
  Time after start of treatment (months) when 50% of patients are free of disease progression (Median PFS). Per RECISIT v1.1, Progressive Disease: ≥20%increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
6-month Progression-free Survival (PFS) | At 6 months
  Proportion of patients alive at 6 months after start of treatment who did not experience disease progression. Per RECISIT v1.1, Progressive Disease: ≥20%increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
Overall Survival (OS) | Up to 40 months
  Time after start of treatment (months) when 50% of patients are alive (Median OS).
6-month Overall Survival (OS) | At 6 months
  Proportion of patients alive at 6 months after start of treatment.
12-month Overall Survival (OS) | At 12 months
  Proportion of patients alive at 12 months after start of treatment.
24-month Overall Survival (OS) | At 24 months
  Proportion of patients alive at 24 months after start of treatment.
36-month Overall Survival (OS) | At 36 months
  Proportion of patients alive at 36 months after start of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Anwaar M Saeed, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (3):
- United States (3):
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Houston Methodist Neal Cancer Center, Houston, Texas
  - Mays Cancer Center, UT Health San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No